CLINICAL TRIAL: NCT03535831
Title: Princess Margaret Cancer Centre 18F-DCFPyL PET Registry
Brief Title: PSMA PET Registry (18F-DCFPyL)
Acronym: PM-PPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-6021
Record Dates: First submitted 2018-04-21; First posted 2018-05-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma of Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single arm study to assess the contribution of 18F-DCFPyL PET imaging (PET/MR or PET/CT) to the management of patients with prostate cancer (PCa).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL PET/ MR or PET/CT imaging (Experimental): Will use a newer technology called PET-MR that combines a Positron Emission Tomography (PET) scan with Magnetic Resonance Imaging (MRI) scan. This new combined imaging test, where PET and MRI data is gathered at one time, will be performed on an integrated PET-MR scanner located at Toronto General Hospital.
  Or technology called PET-CT that combines a Positron Emission Tomography (PET) scan with a computed tomography (CT) scan. This combined imaging test, where PET and CT data is gathered at one time, will be performed on an integrated PET-CT scanner located at Princess Margaret Cancer Centre.
  Choice of imaging method (PET/CT or PET/MR) will be made by one of the study PIs, based on clinical judgement taking into account the specific exam indication, prior recent imaging, and suitability for MR imaging.
  Interventions: Diagnostic Test: 18F-DCFPyL

INTERVENTIONS:
Diagnostic Test: 18F-DCFPyL — The purpose of this study is to determine if use of 18F-DCFPyL would increase the detection of lesions and to better inform your oncologist on the best method of treatment for your disease.

SUMMARY:
The purpose of the Princess Margaret Cancer Centre PSMA registry is to assess the contribution of 18F-DCFPyL (PSMA) PET imaging (PET/MR or PET/CT) to the management of patients with prostate cancer (PCa).

Background:

Currently, patients with intermediate or high risk prostate cancer are staged with CT abdomen and pelvis and bone scan to assess for distant metastases. Patients with biochemical recurrence after primary therapy are restaged in a similar manner. Locally, multiparametric MR of the prostate or prostate bed may also be obtained in select cases.

Patients recruited for this registry will be staged/ restaged with PSMA PET (PET/CT or PET/MR) to determine whether this imaging strategy results in more accurate detection of metastatic disease (for patients undergoing primary staging) or detection of local recurrence or distant disease (for patients undergoing restaging). Choice of imaging method (PET/CT or PET/MR) will be made by one of the study PIs, based on clinical judgement taking into account the specific exam indication, prior recent imaging, and suitability for MR imaging.

Study design:

This is a single arm study to assess the contribution of PSMA PET imaging (PET/MR or PET/CT) to the management of patients with prostate cancer (PCa).

In this prospective trial, the investigators will recruit 200 men whom will undergo PET imaging using an integrated PET/CT scanner or with an integrated PET/MR.

Patients will receive standard treatment for PCa according to UHN/PMH urology oncology site policies.

Treatment outcome including clinical response, blood work including serial serum PSA, and follow-up imaging if performed up to 5 years will be recorded.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most common cancer among Canadian men. Men diagnosed with localized PCa are placed in low, intermediate and high-risk groups, using the prognostic variables including pathologic Gleason score, T-stage and serum prostate specific antigen (PSA). These risk groups correlate with biochemical failure-free survival and prostate cancer specific mortality [1]. Although PCa is prevalent, the risk of clinical or fatal PCa in a 50 year old man is estimated at only 10% and 3%, respectively [2]. Currently, over 2/3 of men diagnosed with PCa are diagnosed with organ confined, low risk disease (PSA < 10 ng/ml, Gleason score (=GS) 3+3, cT1c) [3]. Management is dependent on tumor grade, size and stage and clinical parameters (e.g. life expectancy) and may range from active surveillance to radical therapy including definitive whole gland treatment (radical prostatectomy (RP), or radiotherapy). Although radical whole gland therapy is effective from an oncological standpoint, it may be associated with significant side effects. A more conservative approach in select patients may be enrollment in an active surveillance program. The concept behind this approach is that small volume, low grade PCa may have an indolent course and may not progress to biological significance in the absence of treatment in the patient's lifetime.

Rationale for this study is to determine in a prospective cohort of patients with unfavorable intermediate-risk or high-risk PCa, whether PSMA PET improves the detection of lymph node and distant metastases as compared to conventional imaging strategies (CT abdomen and bone scintigraphy).

To determine the rate of change in planned management after adding information from PSMA PET in patients with PCa being staged prior to primary therapy or restaged after primary therapy.

The central hypothesis behind the Princess Margaret Cancer Centre PSMA PET registry is that in patients with PCa, PSMA PET will enable more accurate staging and restaging, and improve prognostic stratification as compared to conventional workup. Furthermore, the investigators hypothesize that the addition of PSMA PET to the workup of these patients will change the planned management in a significant proportion of patients.

Primary Objective:

To determine in a prospective cohort of patients with unfavorable intermediate-risk or high-risk PCa, whether PSMA PET improves the detection of lymph node and distant metastases as compared to conventional imaging strategies (CT abdomen and bone scintigraphy).

To determine the rate of change in planned management after adding information from PSMA PET in patients with PCa being staged prior to primary therapy or restaged after primary therapy.

Secondary Objective:

To determine the clinical outcome and rate of biochemical control after therapy. For this purpose, information from clinical notes of routine clinical visits, results of blood tests (such as serum PSA) and follow-up imaging, if performed, will be collected for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion in this study if they meet all of the following criteria:
* Age ≥ 18 years
* Histologic diagnosis of carcinoma of prostate
* Being staged or restaged for any of the following indications:

A. Staging of patients with:

i. High risk disease; defined as at least one of the following: a. Gleason ≥8, b. ≥T3 disease, c. PSA >20 ng/ml; ii. Unfavourable intermediate-risk disease defined as: a. more than one intermediate-risk factor (cT2b/ cT2c; GS=7; serum PSA of 10-20 ng/ml); or b. Gleason score of 4+3=7 or more; or c. greater than 50% positive biopsy cores.

B. Staging or restaging of PCa with equivocal findings on conventional workup:

i. Patients with PCa being staged or restaged with equivocal findings on conventional workup (CT, bone scan, MRI); to help guide management or select appropriate site for biopsy to establish disease status.

C. Restaging of patients with:

i. Biochemical failure (BCF) after primary therapy (radical prostatectomy or primary radiotherapy), or ii. BCF after salvage therapy/therapies when further treatment is being considered or iii. Pathologically involved nodes at time of radical prostatectomy or iv. Persistently detectable PSA (>0.1 ng/ml) >3 months after prostatectomy 5.1.4 Ability to provide written informed consent to participate in the study

Exclusion Criteria:

* Patients will be ineligible to participate in this study if they meet any of the following criteria:
* Inability to lie still for PET/CT or PET/MR examination
* For patients undergoing PET/MR only, any contraindication to MRI as per Joint Department of Medical Imaging policies (this exclusion criterion would not exclude patient from enrolling in the registry and undergoing PET/CT).
* Patients with documented, clear-cut metastatic disease on conventional workup where PET findings would not potentially alter patient management. In case of uncertainty, the patient will be discussed at multidisciplinary tumor boards and a majority decision will be made

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
18F-DCFPyL PET changes the detection of lymph node and distant metastases | Through study completion up to 5 years
  To determine in a prospective cohort of patients with unfavorable intermediate-risk or high-risk PCa, whether 18F-DCFPyL PET improves the detection of lymph node and distant metastases as compared to conventional imaging strategies (CT abdomen and bone scintigraphy).

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mirshahvalad SA, Basso Dias A, Ortega C, Abreu Gomez JA, Krishna S, Perlis N, Berlin A, van der Kwast T, Jhaveri K, Ghai S, Metser U, Santiago AT, Veit-Haibach P. [18F]F-DCFPyL PET/MRI radiomics for intraprostatic prostate cancer detection and metastases prediction using whole-gland segmentation. Br J Radiol. 2025 Oct 1;98(1174):1606-1614. doi: 10.1093/bjr/tqaf014. PMID 39847533
- [Derived] Basso Dias A, Finelli A, Bauman G, Veit-Haibach P, Berlin A, Ortega C, Avery L, Metser U. Impact of 18F-DCFPyL PET on Staging and Treatment of Unfavorable Intermediate or High-Risk Prostate Cancer. Radiology. 2022 Sep;304(3):600-608. doi: 10.1148/radiol.211836. Epub 2022 May 24. PMID 35608445